CLINICAL TRIAL: NCT04168190
Title: A Phase 1/Phase 2, Randomized, Double-blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Polyvalent Pneumococcal Conjugate Vaccine in Adults.
Brief Title: A Phase 1/Phase 2 Study of Polyvalent Pneumococcal Conjugate Vaccine (V116) in Adults (V116-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: pPCV-001; pPCV-001 (Other: Merck Protocol Number); V116-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2019-11-18; First posted 2019-11-19 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: V116 0.5 mL (Experimental): Participants will receive a single intramuscular (IM) 0.5 mL vaccination on Day 1 of Phase 1
  Interventions: Biological: V116
- Phase 1: V116 1.0 mL (Experimental): Participants will receive a single IM 1.0 mL vaccination on Day 1 of Phase 1
  Interventions: Biological: V116
- Phase 1: Pneumovax™23 (Active Comparator): Participants will receive a single IM 0.5 mL vaccination on Day 1 of Phase 1
  Interventions: Biological: Pneumovax™23
- Phase 2: V116 (Experimental): Participants will receive a single IM 1.0 mL vaccination on Day 1 of Phase 2
  Interventions: Biological: V116
- Phase 2: Pneumovax™23 (Active Comparator): Participants will receive a single IM 0.5 mL vaccination on Day 1 of Phase 2
  Interventions: Biological: Pneumovax™23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 2 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Polyvalent pneumococcal conjugate vaccine (pPCV); Pneumococcal 21-valent Conjugate Vaccine
  Arms: Phase 1: V116 0.5 mL; Phase 1: V116 1.0 mL; Phase 2: V116
Biological: Pneumovax™23 — Pneumococcal 23-valent polyvalent vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PPSV23
  Arms: Phase 1: Pneumovax™23; Phase 2: Pneumovax™23

SUMMARY:
This Phase 1 and Phase 2 study will evaluate the safety, tolerability and immunogenicity of V116 when administered to adults. Phase 1 has no formal hypothesis. The primary hypotheses for Phase 2 are: V116 is noninferior to Pneumovax™23 as measured by the serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) for the common serotypes at 30 days postvaccination and that the serotype-specific OPA GMTs for the unique serotypes in V116 at 30 days postvaccination are statistically significantly greater following vaccination with V116 than those following vaccination with Pneumovax™23.

ELIGIBILITY:
Inclusion Criteria

* Phase 1:
* Male or female, from 18 years to 49 years of age inclusive
* Phase 2:
* Male or female ≥50 years of age Phase 1 and Phase 2
* Males: refrain from donating sperm, remain abstinent during study or agree to use condom
* Females: Not pregnant. If a woman of childbearing potential, agree to use contraception or remain abstinent

Exclusion Criteria

* History of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease within 3 years of screening
* Known hypersensitivity to any component of the pPCV, or any diphtheria toxoid-containing vaccine
* Known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease
* Coagulation disorder contraindicating IM vaccination
* Recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring within 72 hours of screening
* Known malignancy that is progressing or has required active treatment within 3 years.(Note: participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [eg, breast carcinoma, cervical cancer in situ] that have undergone potentially curative therapy are not excluded)
* Pregnant
* Received any pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study, outside of the protocol.
* Receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received a blood transfusion or blood products, including immunoglobulin, 6 months before study vaccination or is scheduled to receive a blood transfusion or blood product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (20):
- United States (20):
  - Simon Williamson Clinic ( Site 0004), Birmingham, Alabama
  - Central Arizona Medical Associates ( Site 0003), Mesa, Arizona
  - Clinical Research of South Florida ( Site 0008), Coral Gables, Florida
  - Indago Research & Health Center, Inc ( Site 0011), Hialeah, Florida
  - Research Centers of America, LLC ( Site 0001), Hollywood, Florida
  - QPS Miami Research Associates ( Site 0016), Miami, Florida
  - L&C Professional Medical Research Institute ( Site 0009), Miami, Florida
  - Advanced Medical Research Institute ( Site 0010), Miami, Florida
  - Optimal Research ( Site 0006), Peoria, Illinois
  - Benchmark Research ( Site 0012), Metairie, Louisiana
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0018), Troy, Michigan
  - Meridian Clinical Research, LLC ( Site 0024), Norfolk, Nebraska
  - Wake Research Clinical Research Center of Nevada, LLC ( Site 0014), Las Vegas, Nevada
  - Meridian Clinical Research, LLC ( Site 0025), Endwell, New York
  - Rochester Clinical Research, Inc. ( Site 0002), Rochester, New York
  - PriMED Clinical Research ( Site 0021), Dayton, Ohio
  - Advanced Medical Research ( Site 0017), Maumee, Ohio
  - Kaiser Permanente Center for Health Research ( Site 0015), Portland, Oregon
  - Diagnostics Research Group ( Site 0013), San Antonio, Texas
  - Advanced Clinical Research ( Site 0022), West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Platt H, Omole T, Cardona J, Fraser NJ, Mularski RA, Andrews C, Daboul N, Gallagher N, Sapre A, Li J, Polis A, Fernsler D, Tamms G, Xu W, Murphy R, Skinner J, Joyce J, Musey L. Safety, tolerability, and immunogenicity of a 21-valent pneumococcal conjugate vaccine, V116, in healthy adults: phase 1/2, randomised, double-blind, active comparator-controlled, multicentre, US-based trial. Lancet Infect Dis. 2023 Feb;23(2):233-246. doi: 10.1016/S1473-3099(22)00526-6. Epub 2022 Sep 15. PMID 36116461

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: V116 0.5 mL: Participants received a single intramuscular (IM) 0.5 mL vaccination on Day 1 of Phase 1
- Phase 1: V116 1.0 mL: Participants received a single IM 1.0 mL vaccination on Day 1 of Phase 1
- Phase 1: Pneumovax™23: Participants received a single IM 0.5 mL vaccination on Day 1 of Phase 1
- Phase 2: V116: Participants received a single IM 1.0 mL vaccination on Day 1 of Phase 2
- Phase 2: Pneumovax™23: Participants received a single IM 0.5 mL vaccination on Day 1 of Phase 2
Period: Overall Study
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23 | Phase 2: V116 | Phase 2: Pneumovax™23
Started | 30 | 30 | 30 | 254 | 256
Treated | 30 | 30 | 30 | 254 | 254
Completed | 29 | 29 | 30 | 244 | 247
Not Completed | 1 | 1 | 0 | 10 | 9
Not completed — Lost to Follow-up | 0 | 1 | 0 | 7 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 4
Not completed — Death | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23 | Phase 2: V116 | Phase 2: Pneumovax™23 | Total
Number analyzed (Participants) | 30 | 30 | 30 | 254 | 256 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (7.4) | 34.7 (8.9) | 35.2 (8.2) | 61.3 (7.0) | 61.2 (7.3) | 57.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 24 | 142 | 140 | 341
  Male | 14 | 11 | 6 | 112 | 116 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 13 | 107 | 107 | 254
  Not Hispanic or Latino | 16 | 17 | 17 | 147 | 147 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 1 | 3
  Asian | 1 | 1 | 2 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 6 | 4 | 4 | 25 | 30 | 69
  White | 23 | 23 | 24 | 224 | 220 | 514
  More than one race | 0 | 2 | 0 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Injection-site AEs solicited on the Vaccine Report Card (VRC) were redness/erythema, swelling, and tenderness/pain. The percentage of participants with one or more solicited injection-site AE was assessed.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants enrolled in Phase 1 portion who received study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants
  Injection site erythema | 10.0 | 23.3 | 20.0
  Injection site pain | 73.3 | 76.7 | 56.7
  Injection site swelling | 20.0 | 16.7 | 13.3
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Injection site erythema; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = -10.0, 95% CI 2-sided [-29.3 to 9.0] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Injection site erythema; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.3, 95% CI 2-sided [-18.1 to 24.6] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Injection site pain; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 16.7, 95% CI 2-sided [-7.7 to 39.3] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Injection site pain; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 20.0, 95% CI 2-sided [-4.1 to 42.1] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Injection site swelling; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 6.7, 95% CI 2-sided [-13.2 to 26.5] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Injection site swelling; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.3, 95% CI 2-sided [-16.0 to 22.8] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23

2. Primary Outcome: Phase 1: Percentage of Participants With a Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Systemic AEs solicited on the VRC were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. The percentage of participants with one or more solicited systemic AE was assessed.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants enrolled in Phase 1 portion who received study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants
  Fatigue | 26.7 | 26.7 | 16.7
  Arthralgia | 16.7 | 10.0 | 6.7
  Myalgia | 26.7 | 30.0 | 13.3
  Headache | 30.0 | 20.0 | 16.7
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Fatigue; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 10.0, 95% CI 2-sided [-11.4 to 31.0] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Fatigue; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 10.0, 95% CI 2-sided [-11.4 to 31.0] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Arthralgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 10.0, 95% CI 2-sided [-7.4 to 28.3] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Arthralgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.3, 95% CI 2-sided [-13.1 to 20.2] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Myalgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 13.3, 95% CI 2-sided [-7.5 to 33.8] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Myalgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 16.7, 95% CI 2-sided [-4.6 to 37.3] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Headache; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 13.3, 95% CI 2-sided [-8.5 to 34.5] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Headache; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.3, 95% CI 2-sided [-17.2 to 23.8] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23

3. Primary Outcome: Phase 1: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with one or more SAE that were assessed by the investigator to be at least possibly related to the study vaccination were reported.
Time Frame: Up to Day 195
Population: All randomized participants enrolled in Phase 1 portion who received study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-11.5 to 11.5] — Phase 1: V116 0.5 mL minus Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-11.5 to 11.5] — Phase 1: V116 1.0 mL minus Phase 1: Pneumovax™23

4. Primary Outcome: Phase 2: Percentage of Participants With a Solicited Injection-site AE
Description: as for outcome 1
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants enrolled in Phase 2 portion who received study vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 254 | 254
Percentage of Participants
  Injection site erythema | 8.7 | 6.7
  Injection site pain | 46.5 | 37.8
  Injection site swelling | 11.0 | 7.9
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Injection site erythema; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 2.0, 95% CI 2-sided [-2.8 to 6.8] — Phase 2: V116 minus Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Injection site pain; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 8.7, 95% CI 2-sided [0.1 to 17.1] — Phase 2: V116 minus Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Injection site swelling; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.1, 95% CI 2-sided [-2.0 to 8.4] — Phase 2: V116 minus Phase 2: Pneumovax™23

5. Primary Outcome: Phase 2: Percentage of Participants With a Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Systemic AEs solicited on the VRC were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. The percentage of participants with 1 or more solicited systemic AE was assessed.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants enrolled in Phase 2 portion who received study vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 254 | 254
Percentage of Participants
  Fatigue | 19.3 | 12.2
  Arthralgia | 4.3 | 4.3
  Myalgia | 11.0 | 9.4
  Headache | 16.9 | 13.4
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Fatigue; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 7.1, 95% CI 2-sided [0.8 to 13.5] — Phase 2: V116 minus Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Arthralgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-3.8 to 3.8] — Phase 2: V116 minus Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Myalgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 1.6, 95% CI 2-sided [-3.8 to 7.0] — Phase 2: V116 minus Phase 2: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Headache; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 3.5, 95% CI 2-sided [-2.7 to 9.9] — Phase 2: V116 minus Phase 2: Pneumovax™23

6. Primary Outcome: Phase 2: Percentage of Participants With Vaccine-related SAEs
Description: An SAE is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants who experienced at least one SAE that were assessed by the investigator to be at least possibly related to the study vaccination were reported.
Time Frame: Up to Day 293
Population: All randomized participants enrolled in Phase 2 portion who received study vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 254 | 254
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-1.5 to 1.5] — Phase 2: V116 minus Phase 2: Pneumovax™23

7. Primary Outcome: Phase 2: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the Common Serotypes in V116 and Pneumovax™23
Description: GMTs for the serotypes common to V116 and Pneumovax™23 were determined using the muliplex opsonophagocytic assay (MOPA). Serotype-specific OPA GMTs and GMT ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) model. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days post vaccination
Population: All randomized participants enrolled in Phase 2 portion without deviations from the protocol that may have substantially affected the results of this immunogenicity endpoint and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 252 | 254
Titers
  Serotype 3 | 226.26 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 226.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 3535.44 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2906.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 2388.12 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2116.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 8213.56 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5192.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 28129.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 29974.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 1504.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1526.78 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 10327.15 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9106.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 6062.22 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5092.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 2840.38 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1252.27 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 2549.45 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 991.10 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 18394.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11249.90 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 9305.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5068.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 3. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — Non-inferiority can be concluded if the lower bound of the 95% CI for the estimated GMT ratio (V116/PPSV23) is >0.33 (1-sided p-value <0.025); p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.00, 95% CI 2-sided [0.82 to 1.22] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 7F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.22, 95% CI 2-sided [0.95 to 1.56] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 19A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.13, 95% CI 2-sided [0.90 to 1.41] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 22F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.58, 95% CI 2-sided [1.16 to 2.16] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 33F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 0.94, 95% CI 2-sided [0.71 to 1.24] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 8. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 0.99, 95% CI 2-sided [0.80 to 1.21] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 9N. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.13, 95% CI 2-sided [0.87 to 1.47] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 10A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.19, 95% CI 2-sided [0.93 to 1.52] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 11A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 2.27, 95% CI 2-sided [1.78 to 2.90] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 12F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 2.57, 95% CI 2-sided [1.86 to 3.55] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 17F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.64, 95% CI 2-sided [1.24 to 2.16] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 20A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 1.84, 95% CI 2-sided [1.43 to 2.36] — Phase 2: V116/Phase 2: Pneumovax™23

8. Primary Outcome: Phase 2: Serotype-specific OPA GMTs for the Unique Serotypes in V116
Description: GMTs for the serotypes unique to V116 were determined using the MOPA. Serotype-specific OPA GMTs and GMT ratios with 95% CIs were calculated using a cLDA model. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days post vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 252 | 254
Titers
  Serotype 6A | 2757.55 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 456.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 11640.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1711.40 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 12611.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4200.74 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 9820.72 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 539.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 11554.45 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 593.91 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 3137.15 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 105.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 7640.78 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 238.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 4461.98 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 127.84 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B | 15704.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1745.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 6A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — Superiority can be concluded if the lower bound of the 95% CI for the estimated GMT ratio (V116/PPSV23) is >1.0 (1-sided p-value <0.025); p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 6.03, 95% CI 2-sided [4.23 to 8.62] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 15A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 6.80, 95% CI 2-sided [5.37 to 8.62] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 15C. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 3.00, 95% CI 2-sided [2.31 to 3.90] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 16F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 18.21, 95% CI 2-sided [12.98 to 25.57] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 23A. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 19.45, 95% CI 2-sided [12.87 to 29.40] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 23B. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 29.88, 95% CI 2-sided [20.72 to 43.09] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 24F. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 32.02, 95% CI 2-sided [22.83 to 44.89] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 31. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 34.90, 95% CI 2-sided [24.25 to 50.23] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 35B. Geometric mean titer (GMT) ratio and 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMT Ratio = 9.00, 95% CI 2-sided [7.19 to 11.26] — Phase 2: V116/Phase 2: Pneumovax™23

9. Secondary Outcome: Phase 1: Serotype-specific Immunoglobin G (IgG) Geometric Mean Concentrations (GMCs) for the Common Serotypes in V116 and Pneumovax™23
Description: Serotype-specific pneumococcal IgG antibodies were measured using pneumococcal electrochemiluminescence (PnECL). Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% confidence intervals were calculated using a cLDA model. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days post vaccination
Population: All randomized participants enrolled in Phase 1 portion without deviations from the protocol that may have substantially affected the results of this immunogenicity endpoint and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
μg/mL
  Serotype 3 | 0.78 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 0.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.86 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 3.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.98 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 6.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10.27 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.93 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 5.27 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 8.64 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 15.19 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11.51 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 11.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17.80 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 5.40 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8.60 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 8.90 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.15 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 4.50 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.44 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.93 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 1.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 11.54 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 15.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 16.44 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 19.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 3; Test type: Other — Geometric mean concentration (GMC) ratio and 95% confidence interval (CI) are estimated from a constrained longitudinal data analysis (cLDA) model; GMC Ratio = 0.91, 95% CI 2-sided [0.58 to 1.42] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 3; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.12, 95% CI 2-sided [0.71 to 1.76] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 7F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.12, 95% CI 2-sided [0.63 to 1.99] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 7F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 2.14, 95% CI 2-sided [1.19 to 3.84] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 19A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.27, 95% CI 2-sided [0.74 to 2.21] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 19A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 2.08, 95% CI 2-sided [1.19 to 3.63] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 22F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.74, 95% CI 2-sided [0.37 to 1.46] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 22F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.00, 95% CI 2-sided [0.50 to 2.00] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 33F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.75, 95% CI 2-sided [0.40 to 1.41] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 33F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.32, 95% CI 2-sided [0.70 to 2.48] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 8; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.64, 95% CI 2-sided [0.37 to 1.08] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 8; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.99, 95% CI 2-sided [0.58 to 1.69] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 13: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 9N; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.03, 95% CI 2-sided [0.57 to 1.85] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 14: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 9N; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.64, 95% CI 2-sided [0.90 to 2.97] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 15: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 10A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.25, 95% CI 2-sided [0.67 to 2.32] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 16: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 10A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.84, 95% CI 2-sided [0.98 to 3.45] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 17: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 11A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.76, 95% CI 2-sided [0.42 to 1.38] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 18: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 11A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.59, 95% CI 2-sided [0.87 to 2.91] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 19: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 12F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.04, 95% CI 2-sided [0.50 to 2.17] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 20: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 12F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 2.14, 95% CI 2-sided [1.02 to 4.50] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 21: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 17F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 2.11, 95% CI 2-sided [1.21 to 3.68] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 22: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 17F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 2.87, 95% CI 2-sided [1.64 to 5.03] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 23: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 20A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.65, 95% CI 2-sided [0.93 to 2.93] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 24: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 20A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.92, 95% CI 2-sided [1.07 to 3.43] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23

10. Secondary Outcome: Phase 1: Serotype-specific Immunoglobin G (IgG) Geometric Mean Concentrations (GMCs) for the Serotypes Unique to V116
Description: Serotype-specific pneumococcal IgG antibodies were measured using PnECL. Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% confidence intervals were calculated using a cLDA model. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days post vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
μg/mL
  Serotype 6A | 6.32 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 8.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.47 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 8.87 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 15.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 16.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 18.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 1.27 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.44 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.37 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 4.02 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 5.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.67 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.61 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 3.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.79 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.42 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 2.68 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35 | 11.89 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 16.09 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 6A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 4.29, 95% CI 2-sided [1.99 to 9.25] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 6A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 5.49, 95% CI 2-sided [2.53 to 11.91] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 15A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 5.05, 95% CI 2-sided [2.59 to 9.85] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 15A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 8.92, 95% CI 2-sided [4.55 to 17.50] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 15C; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 4.40, 95% CI 2-sided [2.38 to 8.15] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 15C; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 4.92, 95% CI 2-sided [2.64 to 9.16] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 16F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 3.41, 95% CI 2-sided [1.97 to 5.91] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 16F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 6.58, 95% CI 2-sided [3.78 to 11.45] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 23A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 9.42, 95% CI 2-sided [4.35 to 20.40] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 23A; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 9.46, 95% CI 2-sided [4.34 to 20.62] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 23B; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 3.43, 95% CI 2-sided [1.95 to 6.05] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 23B; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 4.77, 95% CI 2-sided [2.69 to 8.45] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 13: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 24F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 8.06, 95% CI 2-sided [3.36 to 19.35] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 14: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 24F; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 16.14, 95% CI 2-sided [6.68 to 39.01] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 15: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 31; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 9.14, 95% CI 2-sided [4.93 to 16.95] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 16: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 31; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 13.58, 95% CI 2-sided [7.28 to 25.32] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 17: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 35B; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 9.24, 95% CI 2-sided [5.56 to 15.36] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 18: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 35B; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 12.50, 95% CI 2-sided [7.49 to 20.87] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23

11. Secondary Outcome: Phase 1: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the Common Serotypes in V116 and Pneumovax™23
Description: GMTs for the serotypes common to V116 and Pneumovax™23 were determined using the MOPA. Serotype-specific OPA GMTs and GMT ratios with 95% confidence intervals were calculated using a cLDA model. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days post vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
Titers
  Serotype 3 | 242.35 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 259.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 243.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 4503.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5672.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5122.36 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 3312.61 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4595.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3475.22 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 21336.23 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 26003.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 12905.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 62540.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 137389.68 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 72703.24 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 1830.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2321.18 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2598.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 28204.72 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 26659.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 24483.35 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 10338.92 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 12377.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6623.80 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 2531.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3152.05 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2836.72 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 5171.95 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7279.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3036.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 48838.60 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 51152.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 24816.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 13910.60 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17799.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11430.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 3; Test type: Other — Geometric mean titer (GMT) ratio and 95% confidence interval (CI) are estimated from a constrained longitudinal data analysis (cLDA) model; GMT Ratio = 0.99, 95% CI 2-sided [0.67 to 1.47] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 3; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.06, 95% CI 2-sided [0.72 to 1.57] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 7F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.88, 95% CI [0.54 to 1.42] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 7F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.11, 95% CI 2-sided [0.68 to 1.80] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 19A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.59 to 1.54] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 19A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.32, 95% CI 2-sided [0.81 to 2.15] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 22F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.65, 95% CI 2-sided [0.85 to 3.23] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 22F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 2.01, 95% CI 2-sided [1.03 to 3.96] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 33F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.86, 95% CI 2-sided [0.44 to 1.67] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 33F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.89, 95% CI 2-sided [0.97 to 3.69] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 8; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.70, 95% CI 2-sided [0.46 to 1.08] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 8; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.89, 95% CI 2-sided [0.58 to 1.38] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 13: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 9N; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [0.62 to 2.15] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 14: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 9N; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.09, 95% CI 2-sided [0.58 to 2.04] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 15: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 10A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.56, 95% CI 2-sided [0.90 to 2.71] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 16: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 10A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.87, 95% CI 2-sided [1.08 to 3.23] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 17: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 11A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 0.89, 95% CI 2-sided [0.53 to 1.49] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 18: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 11A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.11, 95% CI 2-sided [0.66 to 1.87] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 19: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 12F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.70, 95% CI 2-sided [0.89 to 3.27] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 20: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 12F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 2.40, 95% CI 2-sided [1.24 to 4.62] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 21: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 17F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.97, 95% CI 2-sided [1.16 to 3.34] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 22: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 17F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 2.06, 95% CI 2-sided [1.21 to 3.51] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 23: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 20A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.22, 95% CI 2-sided [0.77 to 1.91] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 24: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 20A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 1.56, 95% CI 2-sided [0.99 to 2.45] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23

12. Secondary Outcome: Phase 1: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the Unique Serotypes in V116 and Pneumovax™23
Description: as for outcome 11
Time Frame: 30 days post vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
Titers
  Serotype 6A | 7182.41 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 7407.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 513.88 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 19337.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 24580.49 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2615.98 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 20743.02 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 27242.11 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9728.58 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 11120.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17201.69 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2931.40 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 26267.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 36793.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1908.80 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 5258.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8684.75 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 220.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 7593.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11867.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 381.95 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 7417.79 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7453.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 128.36 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B | 21103.18 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 23826.47 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3044.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 6A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 13.98, 95% CI 2-sided [5.90 to 33.10] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 6A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 14.42, 95% CI 2-sided [6.05 to 34.35] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 15A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 7.39, 95% CI [4.29 to 12.75] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 15A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 9.40, 95% CI 2-sided [5.42 to 16.28] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 15C; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 2.13, 95% CI 2-sided [1.25 to 3.63] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 15C; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 2.80, 95% CI 2-sided [1.64 to 4.79] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 16F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 3.79, 95% CI 2-sided [1.88 to 7.67] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 16F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 5.87, 95% CI 2-sided [2.88 to 11.94] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 23A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 13.76, 95% CI 2-sided [5.68 to 33.32] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 23A; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 19.28, 95% CI 2-sided [7.91 to 47.00] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 23B; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 23.85, 95% CI 2-sided [8.64 to 65.82] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 23B; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 39.39, 95% CI 2-sided [14.15 to 109.65] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 13: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 24F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 19.88, 95% CI 2-sided [9.03 to 43.74] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 14: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 24F; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 31.07, 95% CI 2-sided [13.98 to 69.03] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 15: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 31; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 57.79, 95% CI 2-sided [25.15 to 132.78] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 16: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 31; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 58.07, 95% CI 2-sided [25.10 to 134.33] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23
Statistical Analysis 17: Comparison: Phase 1: V116 0.5 mL vs Phase 1: Pneumovax™23; Serotype 35B; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 6.93, 95% CI 2-sided [4.45 to 10.80] — Phase 1: V116 0.5 mL/Phase 1: Pneumovax™23
Statistical Analysis 18: Comparison: Phase 1: V116 1.0 mL vs Phase 1: Pneumovax™23; Serotype 35B; Test type: Other — [test comment as in outcome 11, analysis 1]; GMT Ratio = 7.82, 95% CI 2-sided [5.00 to 12.24] — Phase 1: V116 1.0 mL/Phase 1: Pneumovax™23

13. Secondary Outcome: Phase 1: Geometric Mean Fold Rise (GMFR) From Baseline in GMTs of Serotype-specific OPA
Description: GMTs for the serotypes in V116 and Pneumovax™23 were determined using the MOPA at baseline and 30 days post vaccination and derived from a cLDA model. The GMFR (Day 30 GMT/Day 1 GMT) from baseline (Day 1) to Day 30 of each pneumococcal IgG serotype was calculated.
Time Frame: Baseline (Day 1) and 30 days postvaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
Ratio
  Serotype 3 | 12.90 [8.95 to 18.59] | 10.68 [6.27 to 18.18] | 10.01 [6.62 to 15.14]
  Serotype 7F: number analyzed (Participants) | 30 | 29 | 29
  Serotype 7F | 15.64 [6.94 to 35.23] | 19.68 [9.96 to 38.87] | 34.18 [15.67 to 74.56]
  Serotype 19A | 12.26 [7.03 to 21.38] | 18.34 [10.32 to 32.60] | 14.92 [7.84 to 28.42]
  Serotype 22F: number analyzed (Participants) | 29 | 29 | 29
  Serotype 22F | 92.21 [38.88 to 218.70] | 81.76 [32.42 to 206.23] | 32.64 [14.59 to 73.04]
  Serotype 33F | 17.68 [10.86 to 28.78] | 34.83 [21.63 to 56.09] | 20.24 [11.07 to 37.02]
  Serotype 8 | 39.67 [21.83 to 72.09] | 50.01 [25.73 to 97.20] | 72.24 [38.21 to 136.59]
  Serotype 9N: number analyzed (Participants) | 30 | 28 | 30
  Serotype 9N | 22.91 [10.93 to 48.00] | 19.80 [8.34 to 47.04] | 27.38 [13.87 to 54.03]
  Serotype 10A: number analyzed (Participants) | 26 | 29 | 27
  Serotype 10A | 12.69 [5.39 to 29.87] | 18.21 [8.76 to 37.85] | 10.35 [5.00 to 21.41]
  Serotype 11A | 7.46 [3.40 to 16.39] | 8.23 [4.46 to 15.21] | 7.64 [4.20 to 13.93]
  Serotype 12F: number analyzed (Participants) | 30 | 29 | 29
  Serotype 12F | 360.69 [192.76 to 674.93] | 448.73 [243.29 to 827.65] | 162.71 [85.83 to 308.43]
  Serotype 17F: number analyzed (Participants) | 30 | 28 | 30
  Serotype 17F | 36.57 [17.73 to 75.45] | 37.33 [20.19 to 69.04] | 20.54 [11.70 to 36.08]
  Serotype 20A: number analyzed (Participants) | 29 | 29 | 30
  Serotype 20A | 15.67 [8.21 to 29.92] | 19.20 [10.52 to 35.07] | 14.91 [8.60 to 25.83]
  Serotype 6A: number analyzed (Participants) | 29 | 29 | 30
  Serotype 6A | 311.54 [171.83 to 565.18] | 375.42 [194.76 to 723.64] | 20.95 [9.44 to 46.47]
  Serotype 15A: number analyzed (Participants) | 30 | 29 | 29
  Serotype 15A | 31.56 [12.49 to 79.74] | 29.31 [13.47 to 63.79] | 5.53 [2.96 to 10.35]
  Serotype 15C: number analyzed (Participants) | 30 | 27 | 28
  Serotype 15C | 37.97 [13.68 to 105.40] | 58.39 [20.58 to 165.67] | 10.58 [6.14 to 18.23]
  Serotype 16F: number analyzed (Participants) | 29 | 28 | 30
  Serotype 16F | 16.82 [7.30 to 38.75] | 25.99 [10.54 to 64.09] | 4.30 [2.59 to 7.12]
  Serotype 23A: number analyzed (Participants) | 29 | 29 | 30
  Serotype 23A | 380.08 [136.77 to 1056.21] | 269.90 [86.95 to 837.80] | 17.52 [6.87 to 44.65]
  Serotype 23B: number analyzed (Participants) | 30 | 29 | 29
  Serotype 23B | 99.58 [36.09 to 274.72] | 157.02 [61.06 to 403.76] | 5.39 [2.92 to 9.95]
  Serotype 24F: number analyzed (Participants) | 29 | 27 | 30
  Serotype 24F | 14.86 [5.86 to 37.70] | 23.51 [9.64 to 57.34] | 1.24 [0.76 to 2.03]
  Serotype 31: number analyzed (Participants) | 29 | 29 | 30
  Serotype 31 | 95.53 [36.62 to 249.17] | 94.51 [39.26 to 227.50] | 3.23 [1.52 to 6.86]
  Serotype 35B | 13.68 [7.26 to 25.79] | 12.56 [8.48 to 18.61] | 1.73 [1.45 to 2.06]
  Serotype 6C | 41.71 [14.41 to 120.73] | 65.05 [23.86 to 177.35] | 2.82 [1.46 to 5.43]
  Serotype 15B | 78.68 [25.58 to 242.03] | 89.25 [30.60 to 260.27] | 33.11 [13.27 to 82.61]
  Serotype 20B | 3.78 [1.97 to 7.26] | 4.17 [2.05 to 8.47] | 5.01 [2.46 to 10.23]

14. Secondary Outcome: Phase 1: Geometric Mean Fold Rise (GMFR) From Baseline in GMCs of Serotype-specific IgG
Description: GMCs for the serotypes in V116 and Pneumovax™23 were measured by PnECL at baseline and 30 days post vaccination and derived from a cLDA model. The GMFR (Day 30 GMC/Day 1 GMC) from baseline (Day 1) to Day 30 of each pneumococcal IgG serotype was calculated.
Time Frame: Baseline (Day 1) and 30 days post vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: Pneumovax™23
Number analyzed (Participants) | 30 | 29 | 30
Ratio
  Serotype 3 | 5.36 [3.90 to 7.35] | 5.94 [4.05 to 8.71] | 4.97 [3.39 to 7.27]
  Serotype 7F | 8.38 [5.30 to 13.25] | 16.00 [10.28 to 24.90] | 7.44 [5.05 to 10.97]
  Serotype 19A | 4.67 [3.03 to 7.21] | 7.28 [4.63 to 11.45] | 3.66 [2.66 to 5.04]
  Serotype 22F | 19.51 [11.64 to 32.69] | 21.83 [13.51 to 35.29] | 24.34 [12.30 to 48.18]
  Serotype 33F | 9.33 [5.62 to 15.49] | 16.28 [10.36 to 25.58] | 11.75 [7.66 to 18.03]
  Serotype 8 | 13.86 [8.94 to 21.49] | 22.89 [15.29 to 34.27] | 25.99 [15.35 to 44.00]
  Serotype 9N | 12.90 [8.60 to 19.36] | 20.85 [13.11 to 33.16] | 14.37 [8.41 to 24.55]
  Serotype 10A | 11.36 [6.61 to 19.52] | 16.10 [9.76 to 26.57] | 9.58 [6.94 to 13.24]
  Serotype 11A | 2.71 [1.70 to 4.33] | 7.18 [3.96 to 13.02] | 5.17 [3.24 to 8.24]
  Serotype 12F | 10.35 [6.36 to 16.85] | 22.71 [13.35 to 38.61] | 9.75 [5.37 to 17.71]
  Serotype 17F | 19.23 [11.44 to 32.34] | 22.52 [14.61 to 34.73] | 10.07 [6.80 to 14.91]
  Serotype 20A | 10.81 [6.67 to 17.50] | 11.18 [7.38 to 16.93] | 5.60 [3.58 to 8.77]
  Serotype 6A | 23.58 [12.37 to 44.95] | 29.48 [18.01 to 48.26] | 5.66 [3.29 to 9.76]
  Serotype 15A | 14.61 [8.07 to 26.45] | 28.84 [17.91 to 46.44] | 3.02 [1.87 to 4.88]
  Serotype 15C | 31.93 [18.64 to 54.69] | 37.55 [20.18 to 69.88] | 7.94 [5.56 to 11.36]
  Serotype 16F | 4.39 [2.71 to 7.11] | 10.80 [7.22 to 16.15] | 1.69 [1.16 to 2.45]
  Serotype 23A | 23.43 [12.21 to 44.99] | 22.53 [11.84 to 42.86] | 2.75 [1.83 to 4.13]
  Serotype 23B | 9.03 [4.99 to 16.36] | 15.56 [8.88 to 27.27] | 2.66 [1.92 to 3.68]
  Serotype 24F | 11.18 [5.18 to 24.13] | 19.44 [11.30 to 33.47] | 1.26 [0.79 to 2.03]
  Serotype 31 | 12.83 [7.24 to 22.75] | 19.71 [12.90 to 30.13] | 1.77 [1.19 to 2.63]
  Serotype 35B | 9.77 [5.70 to 16.73] | 11.33 [7.01 to 18.31] | 0.96 [0.86 to 1.06]
  Serotype 6C | 6.52 [3.64 to 11.70] | 9.48 [5.47 to 16.42] | 2.22 [1.61 to 3.07]
  Serotype 15B | 12.54 [6.73 to 23.36] | 11.96 [6.32 to 22.65] | 8.05 [5.67 to 11.42]

15. Secondary Outcome: Phase 2: Serotype-specific IgG GMCs for the Common Serotypes in V116 and Pneumovax™23
Description: as for outcome 10
Time Frame: 30 days post vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 252 | 254
μg/mL
  Serotype 3 | 0.78 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 0.72 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 4.98 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 7.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 3.81 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.79 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 11.89 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 9.86 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10.30 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 7.18 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.51 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 10.78 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.89 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 5.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.35 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 1.56 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.68 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 12.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.06 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 20.59 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.09 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 3. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — Non-inferiority can be concluded if the lower bound of the 95% CI for the estimated GMC ratio (V116/PPSV23) is >0.5 (1-sided p-value <0.025); p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.08, 95% CI 2-sided [0.90 to 1.30] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 7F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.23, 95% CI 2-sided [0.99 to 1.52] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 19A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.24, 95% CI 2-sided [1.02 to 1.52] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 22F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.36, 95% CI 2-sided [1.06 to 1.75] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 33F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 0.86, 95% CI 2-sided [0.69 to 1.06] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 8. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 0.96, 95% CI 2-sided [0.78 to 1.18] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 9N. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.30, 95% CI 2-sided [1.04 to 1.64] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 10A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.83, 95% CI 2-sided [1.44 to 2.32] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 11A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.54, 95% CI 2-sided [1.27 to 1.86] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 10: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 12F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 2.30, 95% CI 2-sided [1.75 to 3.04] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 11: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 17F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 1.82, 95% CI 2-sided [1.49 to 2.22] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 12: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 20A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 2.27, 95% CI 2-sided [1.81 to 2.83] — Phase 2: V116/Phase 2: Pneumovax™23

16. Secondary Outcome: Phase 2: Serotype-specific IgG GMCs for the Serotypes Unique to V116
Description: as for outcome 10
Time Frame: 30 days post vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 252 | 254
μg/mL
  Serotype 6A | 4.06 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 1.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 13.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 11.91 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 2.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 3.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.42 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 5.18 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.92 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 6.11 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 3.15 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B | 24.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 6A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — Superiority can be concluded if the lower bound of the 95% CI for the estimated GMC ratio (V116/PPSV23) is >1.0 (1-sided p-value <0.025); p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 3.77, 95% CI 2-sided [2.95 to 4.84] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 2: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 15A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 7.68, 95% CI 2-sided [6.12 to 9.64] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 3: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 15C. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 3.29, 95% CI 2-sided [2.60 to 4.17] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 4: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 16F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 8.65, 95% CI 2-sided [7.19 to 10.41] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 5: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 23A. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 7.83, 95% CI 2-sided [6.20 to 9.90] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 6: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 23B. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 5.61, 95% CI 2-sided [4.53 to 6.94] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 7: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 24F. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 23.99, 95% CI 2-sided [19.35 to 29.74] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 8: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 31. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value was estimated from a cLDA model; GMC Ratio = 10.13, 95% CI 2-sided [8.32 to 12.33] — Phase 2: V116/Phase 2: Pneumovax™23
Statistical Analysis 9: Comparison: Phase 2: V116 vs Phase 2: Pneumovax™23; Serotype 35B. Geometric mean concentration (GMC) ratio, 95% confidence interval (CI), and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.001, P-value is estimated from a cLDA model; GMC Ratio = 18.29, 95% CI 2-sided [15.59 to 21.45] — Phase 2: V116/Phase 2: Pneumovax™23

17. Secondary Outcome: Phase 2: Geometric Mean Fold Rise (GMFR) From Baseline in GMTs of Serotype-specific OPA
Description: GMTs for the serotypes in V116 and Pneumovax™23 were determined using the MOPA at baseline and at 30 days post vaccination and derived from a cLDA model. The GMFR for each pneumococcal IgG serotype was calculated as Day 30 GMT/Day 1 GMT.
Time Frame: Baseline (Day 1) and 30 days post vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 238 | 235
Ratio
  Serotype 3 | 12.03 [10.04 to 14.41] | 10.96 [9.25 to 13.00]
  Serotype 7F: number analyzed (Participants) | 236 | 235
  Serotype 7F | 31.07 [22.87 to 42.22] | 22.52 [17.23 to 29.45]
  Serotype 19A: number analyzed (Participants) | 236 | 234
  Serotype 19A | 13.05 [10.22 to 16.66] | 10.26 [8.31 to 12.67]
  Serotype 22F: number analyzed (Participants) | 235 | 232
  Serotype 22F | 52.66 [37.40 to 74.14] | 46.34 [33.34 to 64.41]
  Serotype 33F: number analyzed (Participants) | 234 | 226
  Serotype 33F | 13.47 [10.47 to 17.32] | 14.04 [11.23 to 17.53]
  Serotype 8: number analyzed (Participants) | 235 | 234
  Serotype 8 | 39.06 [30.34 to 50.28] | 40.06 [31.59 to 50.80]
  Serotype 9N: number analyzed (Participants) | 233 | 229
  Serotype 9N | 33.51 [24.38 to 46.04] | 29.38 [21.67 to 39.82]
  Serotype 10A: number analyzed (Participants) | 182 | 174
  Serotype 10A | 12.34 [8.79 to 17.31] | 8.12 [6.03 to 10.94]
  Serotype 11A: number analyzed (Participants) | 238 | 229
  Serotype 11A | 33.21 [25.13 to 43.88] | 12.29 [9.41 to 16.05]
  Serotype 12F: number analyzed (Participants) | 214 | 222
  Serotype 12F | 150.08 [112.83 to 199.61] | 57.03 [42.59 to 76.35]
  Serotype 17F: number analyzed (Participants) | 237 | 230
  Serotype 17F | 40.71 [30.35 to 54.60] | 25.68 [19.56 to 33.73]
  Serotype 20A | 20.48 [16.11 to 26.02] | 12.16 [9.58 to 15.43]
  Serotype 6A: number analyzed (Participants) | 238 | 233
  Serotype 6A | 79.16 [58.28 to 107.51] | 11.30 [8.42 to 15.16]
  Serotype 15A: number analyzed (Participants) | 216 | 211
  Serotype 15A | 26.66 [20.16 to 35.25] | 3.93 [3.18 to 4.87]
  Serotype 15C: number analyzed (Participants) | 226 | 217
  Serotype 15C | 65.18 [46.91 to 90.58] | 23.73 [16.98 to 33.15]
  Serotype 16F: number analyzed (Participants) | 226 | 215
  Serotype 16F | 56.50 [41.53 to 76.85] | 3.54 [2.61 to 4.81]
  Serotype 23A: number analyzed (Participants) | 210 | 197
  Serotype 23A | 237.14 [166.28 to 338.22] | 10.65 [7.42 to 15.29]
  Serotype 23B: number analyzed (Participants) | 230 | 228
  Serotype 23B | 97.79 [71.94 to 132.92] | 4.62 [3.58 to 5.96]
  Serotype 24F: number analyzed (Participants) | 221 | 203
  Serotype 24F | 48.78 [35.07 to 67.84] | 1.52 [1.18 to 1.97]
  Serotype 31: number analyzed (Participants) | 216 | 209
  Serotype 31 | 92.00 [66.09 to 128.07] | 3.25 [2.51 to 4.21]
  Serotype 35B: number analyzed (Participants) | 228 | 221
  Serotype 35B | 12.41 [10.08 to 15.27] | 1.53 [1.33 to 1.75]
  Serotype 6C: number analyzed (Participants) | 231 | 231
  Serotype 6C | 19.41 [13.65 to 27.61] | 4.24 [3.09 to 5.84]
  Serotype 15B: number analyzed (Participants) | 224 | 223
  Serotype 15B | 24.32 [17.88 to 33.08] | 25.73 [19.14 to 34.58]
  Serotype 20B: number analyzed (Participants) | 231 | 227
  Serotype 20B | 7.21 [5.68 to 9.17] | 5.35 [4.08 to 7.01]

18. Secondary Outcome: Phase 2: GMFR From Baseline in GMCs of Serotype-specific IgG
Description: GMCs for each serotype common in V116 and Pneumovax™23 were measured using PnECL at baseline and 30 days post vaccination and derived from a cLDA model. The GMFR for each pneumococcal IgG serotype was calculated as Day 30 GMC/Day 1 GMC.
Time Frame: Baseline (Day 1) and 30 days post vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 240 | 239
Ratio
  Serotype 3 | 5.23 [4.52 to 6.06] | 4.56 [3.98 to 5.21]
  Serotype 7F | 9.96 [8.40 to 11.81] | 8.28 [7.06 to 9.71]
  Serotype 19A | 5.29 [4.51 to 6.21] | 4.12 [3.60 to 4.71]
  Serotype 22F | 12.45 [10.07 to 15.39] | 9.04 [7.53 to 10.86]
  Serotype 33F | 9.94 [8.26 to 11.97] | 11.63 [9.87 to 13.71]
  Serotype 8 | 14.53 [11.92 to 17.72] | 15.51 [13.06 to 18.40]
  Serotype 9N | 17.77 [14.62 to 21.61] | 11.80 [9.92 to 14.04]
  Serotype 10A | 17.32 [14.41 to 20.82] | 9.29 [7.92 to 10.90]
  Serotype 11A | 7.71 [6.56 to 9.07] | 4.72 [4.12 to 5.41]
  Serotype 12F | 13.72 [11.13 to 16.91] | 6.14 [5.11 to 7.37]
  Serotype 17F | 20.26 [17.03 to 24.11] | 11.11 [9.54 to 12.95]
  Serotype 20A | 14.95 [12.53 to 17.84] | 6.30 [5.41 to 7.33]
  Serotype 6A | 13.35 [10.90 to 16.35] | 3.56 [3.03 to 4.19]
  Serotype 15A | 23.94 [19.89 to 28.81] | 3.02 [2.63 to 3.47]
  Serotype 15C | 22.35 [18.49 to 27.01] | 7.28 [6.17 to 8.60]
  Serotype 16F | 12.42 [10.62 to 14.52] | 1.51 [1.37 to 1.66]
  Serotype 23A | 20.27 [16.82 to 24.43] | 2.66 [2.30 to 3.06]
  Serotype 23B | 13.50 [11.25 to 16.21] | 2.51 [2.21 to 2.85]
  Serotype 24F | 25.20 [20.48 to 31.02] | 1.08 [1.02 to 1.14]
  Serotype 31 | 15.89 [13.47 to 18.76] | 1.62 [1.46 to 1.81]
  Serotype 35B | 18.72 [15.89 to 22.05] | 1.04 [0.98 to 1.10]
  Serotype 6C: number analyzed (Participants) | 234 | 239
  Serotype 6C | 5.78 [4.79 to 6.97] | 1.67 [1.52 to 1.85]
  Serotype 15B | 9.95 [8.28 to 11.95] | 8.87 [7.52 to 10.47]

19. Secondary Outcome: Phase 2: Percentage of Participants Who Achieve a ≥4-fold Increase in Serotype-specific OPA Responses From Prevaccination (Baseline [Day 1]) to 30 Days Post Vaccination
Description: The percentage of participants with ≥4-fold rise from baseline (Day 1) to Day 30 in GMTs of each pneumococcal serotype was calculated. Titer levels were determined by the MOPA and derived from a cLDA model.
Time Frame: Baseline (Day 1) and 30 days post vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: V116 | Phase 2: Pneumovax™23
Number analyzed (Participants) | 238 | 235
Percentage of Participants
  Serotype 3 | 74.8 [68.8 to 80.2] | 75.7 [69.7 to 81.1]
  Serotype 7F: number analyzed (Participants) | 236 | 235
  Serotype 7F | 74.2 [68.1 to 79.6] | 77.0 [71.1 to 82.2]
  Serotype 19A: number analyzed (Participants) | 236 | 234
  Serotype 19A | 66.9 [60.6 to 72.9] | 67.1 [60.7 to 73.1]
  Serotype 22F: number analyzed (Participants) | 235 | 232
  Serotype 22F | 81.3 [75.7 to 86.1] | 79.3 [73.5 to 84.3]
  Serotype 33F: number analyzed (Participants) | 234 | 226
  Serotype 33F | 68.4 [62.0 to 74.3] | 75.7 [69.5 to 81.1]
  Serotype 8: number analyzed (Participants) | 235 | 234
  Serotype 8 | 80.9 [75.2 to 85.7] | 85.5 [80.3 to 89.7]
  Serotype 9N: number analyzed (Participants) | 233 | 229
  Serotype 9N | 77.3 [71.3 to 82.5] | 79.5 [73.7 to 84.5]
  Serotype 10A: number analyzed (Participants) | 182 | 174
  Serotype 10A | 59.9 [52.4 to 67.1] | 55.2 [47.5 to 62.7]
  Serotype 11A: number analyzed (Participants) | 238 | 229
  Serotype 11A | 80.3 [74.6 to 85.1] | 62.9 [56.3 to 69.2]
  Serotype 12F: number analyzed (Participants) | 214 | 222
  Serotype 12F | 90.2 [85.4 to 93.8] | 82.9 [77.3 to 87.6]
  Serotype 17F: number analyzed (Participants) | 237 | 230
  Serotype 17F | 85.2 [80.1 to 89.5] | 80.9 [75.2 to 85.7]
  Serotype 20A | 83.6 [78.3 to 88.1] | 69.4 [63.0 to 75.2]
  Serotype 6A: number analyzed (Participants) | 238 | 233
  Serotype 6A | 83.2 [77.8 to 87.7] | 58.8 [52.2 to 65.2]
  Serotype 15A: number analyzed (Participants) | 216 | 211
  Serotype 15A | 86.6 [81.3 to 90.8] | 39.3 [32.7 to 46.3]
  Serotype 15C: number analyzed (Participants) | 226 | 217
  Serotype 15C | 88.5 [83.6 to 92.3] | 71.0 [64.4 to 76.9]
  Serotype 16F: number analyzed (Participants) | 226 | 215
  Serotype 16F | 85.4 [80.1 to 89.7] | 30.2 [24.2 to 36.8]
  Serotype 23A: number analyzed (Participants) | 210 | 197
  Serotype 23A | 93.3 [89.1 to 96.3] | 48.7 [41.6 to 55.9]
  Serotype 23B: number analyzed (Participants) | 230 | 228
  Serotype 23B | 87.4 [82.4 to 91.4] | 40.4 [33.9 to 47.0]
  Serotype 24F: number analyzed (Participants) | 221 | 203
  Serotype 24F | 82.8 [77.2 to 87.5] | 15.3 [10.6 to 21.0]
  Serotype 31: number analyzed (Participants) | 216 | 209
  Serotype 31 | 86.6 [81.3 to 90.8] | 30.1 [24.0 to 36.9]
  Serotype 35B: number analyzed (Participants) | 228 | 221
  Serotype 35B | 73.2 [67.0 to 78.9] | 11.3 [7.5 to 16.2]
  Serotype 6C: number analyzed (Participants) | 231 | 231
  Serotype 6C | 58.4 [51.8 to 64.9] | 33.8 [27.7 to 40.3]
  Serotype 15B: number analyzed (Participants) | 224 | 223
  Serotype 15B | 71.0 [64.6 to 76.8] | 75.3 [69.1 to 80.8]
  Serotype 20B: number analyzed (Participants) | 231 | 227
  Serotype 20B | 52.8 [46.2 to 59.4] | 44.1 [37.5 to 50.8]

ADVERSE EVENTS:
Time Frame: Up to approximately 195 days post-vaccination for Phase 1 and up to approximately 293 days post-vaccination for Phase 2.
Description: The analysis population for All-Cause Mortality included all randomized participants. The safety analysis population included all randomized participants who received the study vaccination. AEs were reported for participants separately during the Phase 1 (MedDRA 23.0) and Phase 2 (MedDRA 24.0) parts of the study.
Groups:
- Phase 1: PPSV23: Participants received a single IM 0.5 mL vaccination on Day 1 of Phase 1
- Phase 2: PPSV23: Participants received a single IM 0.5 mL vaccination on Day 1 of Phase 2
Arm/Group | Phase 1: V116 0.5 mL | Phase 1: V116 1.0 mL | Phase 1: PPSV23 | Phase 2: V116 | Phase 2: PPSV23
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 1/254 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 4/254 | 3/254
Other Adverse Events (participants affected / at risk) | 23/30 | 24/30 | 21/30 | 159/254 | 133/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: V116 0.5 mL (N=30) | Phase 1: V116 1.0 mL (N=30) | Phase 1: PPSV23 (N=30) | Phase 2: V116 (N=254) | Phase 2: PPSV23 (N=254)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: V116 0.5 mL (N=30) | Phase 1: V116 1.0 mL (N=30) | Phase 1: PPSV23 (N=30) | Phase 2: V116 (N=254) | Phase 2: PPSV23 (N=254)
Fatigue (General disorders) | 8 (8) | 8 (8) | 5 (5) | 50 (50) | 32 (34)
Injection site bruising (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 7 (7) | 6 (6) | 26 (26) | 17 (17)
Injection site pain (General disorders) | 22 (23) | 23 (23) | 17 (17) | 118 (119) | 96 (96)
Injection site swelling (General disorders) | 6 (6) | 5 (5) | 4 (4) | 30 (30) | 20 (20)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2) | 11 (14) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) | 4 (4) | 33 (35) | 26 (28)
Headache (Nervous system disorders) | 10 (10) | 6 (6) | 5 (7) | 47 (59) | 41 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04168190/Prot_SAP_000.pdf